CLINICAL TRIAL: NCT05276219
Title: Vasodilation or Loop-diuretics for Initial Treatment of Pulmonary Edema or Congestion Due to Acute Heart Failure - a Randomized Placebo-controlled Trial
Brief Title: Optimized Treatment of Pulmonary Edema or Congestion
Acronym: Decongest
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Grand (Other)
Collaborators: Zealand University Hospital (Other); Copenhagen University Hospital, Hvidovre (Other); Bispebjerg Hospital (Other)
Responsible Party: Sponsor-Investigator, Johannes Grand, Principal investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08102021_ver2.5; 2022-500035-36-01 (Other: euclinicaltrials.eu)
Record Dates: First submitted 2022-01-31; First posted 2022-03-11 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Edema; Congestive Heart Failure; Acute Heart Failure
Keywords: acute heart failure; Pulmonary edema
MeSH Terms: conditions — Pulmonary Edema; Heart Failure | interventions — Furosemide; Isosorbide Dinitrate

STUDY DESIGN:
Intervention Model Description: Inter-regional collaborative, randomized, placebo-controlled trial with 1:1:1 allocation
  * Boluses of 40 mg furosemide given as soon as possible and repeated up to 10 times by the discretion of the treating physician.
  * Boluses of 3 mg IV isosorbide dinitrate given as soon as possible and repeated up to 10 times by the discretion of the treating physician.
  * Boluses of both 3 mg IV isosorbide dinitrate + of 40 mg furosemide given as soon as possible and repeated up to 10 times by the discretion of the treating physician.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching and identical placebo (saline)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Furosemide only (Active Comparator): • Boluses of 40 mg furosemide given as soon as possible and repeated up to 10 times by the discretion of the treating physician.
  Interventions: Drug: Furosemide Injection
- isosorbide dinitrate (Active Comparator): • Boluses of 3 mg IV isosorbide dinitrate given as soon as possible and repeated up to 10 times by the discretion of the treating physician.
  Interventions: Drug: Isosorbide Dinitrate
- isosorbide dinitrate + furosemide (Active Comparator): • Boluses of both 3 mg IV isosorbide dinitrate + of 40 mg furosemide given as soon as possible and repeated up to 10 times by the discretion of the treating physician.
  Interventions: Drug: Furosemide and isosorbide dinitrate

INTERVENTIONS:
Drug: Furosemide Injection — A diuretic (iv furosemide) strategy for decongestion in acute heart failure
  Arms: Furosemide only
Drug: Isosorbide Dinitrate — Vasodilation (iv isosorbide dinitrate) strategy for decongestion in acute heart failure
  Arms: isosorbide dinitrate
Drug: Furosemide and isosorbide dinitrate — Vasodilation (iv isosorbide dinitrate) strategy for decongestion in acute heart failure AND A diuretic (iv furosemide) strategy for decongestion in acute heart failure
  Arms: isosorbide dinitrate + furosemide

SUMMARY:
Background:

Intravenous (IV) loop-diuretics have been a key component in treating pulmonary edema since the nineteen sixties and has a Class 1 recommendation in the 2021 European Society of Cardiology guidelines for heart failure. Conversely, vasodilation was downgraded in the treatment of acute heart failure due to a lack of trials that compare vasodilation with loop-diuretics in a hyperacute clinical setting. This clinical equipoise will be tested in a trial including patients with pulmonary congestion immediately at hospital admission.

Primary objective:

To determine the superior strategy of loop-diuretics (furosemide), vasodilation (nitrates) or the combination during emergency treatment.

Design: Investigator-initiated, randomized, double-blinded, placebo-controlled trial with 1:1:1 allocation.

Intervention:

Intervention-phase will last 6 hours from study-inclusion, and patients will be allocated to one of three groups:

* Boluses of 40 mg IV furosemide + nitrate-placebo as soon as possible and repeated up to 10 times.
* Boluses of 3 mg IV isosorbide dinitrate + furosemide-placebo as soon as possible.
* Boluses of both 3 mg IV isosorbide dinitrate + of 40 mg as soon as possible.

DETAILED DESCRIPTION:
IV-loop diuretics are a central part of acute treatment of pulmonary edema and is recommended in guidelines (Class 1 recommendation) with a higher recommendation as compared to vasodilation, which was downgraded from Ia to IIb in the 2021 guidelines for heart failure. However, the effects of loop-diuretics alone or in combination with nitrates compared to nitrates alone is unknown and should be investigated in adequately powered prospective trials to optimize acute treatment of these patients.

Trial objective The primary objective is to determine the superior strategy of urgent treatment (starting within 3 hours after hospital-admission) of pulmonary edema. Strategies are: 1. Diuretics (Furosemide), 2. Vasodilation (nitrates), 3. A combination of both furosemide and nitrates. Patient-outcome will be evaluated through the primary endpoint as described elsewhere.

Hypothesis:

Iv nitrates in combination with iv furosemide are superior compared to iv furosemide alone or iv nitrates alone during initial (first 6 hours) in-hospital treatment of pulmonary edema. "Superior" is defined as a significant benefit on the primary outcome.

Study design The study is an investigator-initiated, randomized, placebo-controlled, double-blinded, multicenter, interventional, clinical trial. Following successful completion of screening procedures, patients will be randomized in a 1:1:1 fashion to receive either of the 3 treatments-strategies.

Since patients are in cardio-respiratory and mental stress, informed consent prior to the intervention will be impossible. Instead, a legal guardian will be contacted and asked for consent in addition to next of kind and patients regaining mental ability.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years
2. Acute (within minutes to days) onset or worsening of subjective dyspnea*
3. Systolic blood pressure ≥100 mmHg
4. Oxygen saturation <94% or need of oxygen
5. Signs or suspicion of congestion (peripheral edema, rales, and/or clinical suspicion of congestion) *

   * by the best assessment from a medical doctor. Inclusion must not wait on x-ray or other measures: patients suspected of pulmonary congestion should be included immediately.

Exclusion criteria

1. More than 40 mg IV furosemide within the last three hours before randomization including prehospital treatment.
2. More than 3 hours from hospital-admission to randomization
3. Ongoing ventricular taky- or brady-arrythmias or supraventricular arrhythmias with HR > 180 or < 40 bpm.
4. Suspected severe infection or sepsis.

Exclusion criteria are purposely liberal, so patients can be included in accordance with everyday clinical practice. However, a safety criterion will be implemented:

If blood pressure drops below 90 mmHg in 2 measurements with 5 minutes apart and/or if urine production is below 50 ml after 1 hour, the intervention will be stopped, and patients can receive furosemide and nitrates freely.

We purposely chose not to exclude patients with aortic stenosis, since observational studies did not find excess risk of given nitrates to patients with pulmonary edema and aortic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1104 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Days alive and outside hospital | 30 days
  The primary end point is the number of days alive and out of hospital during the 30-day period after the hospital-visit. The choice of this end point allow capturing the burden of acute heart failure in terms of mortality, hospital length of stay, and early readmission to the hospital. Patients who died before day 30 will be counted as having zero days alive and out of hospital. A return visit to the emergency department was considered as 1 day in the hospital, using the same approach as a recent trial of acute heart failure.

SECONDARY OUTCOMES:
A composite outcome consisting of 1. all-cause mortality, 2. in-hospital worsening heart failure (WHF) or 3. hospital readmission for HF through Day 30. | 30 days
  WHF was defined as progress in signs and/or symptoms of heart failure that lead to an intensification of treatment for heart failure. Such treatment was defined as initiation of mechanical ventilation, renal replacement therapy, vasopressors, inotropes, or mechanical heart failure treatment.
Worsening heart failure until day 30 | 30 days
  WHF was defined as progress in signs and/or symptoms of heart failure that lead to an intensification of treatment for heart failure. Such treatment was defined as initiation of mechanical ventilation, renal replacement therapy, vasopressors, inotropes, or mechanical heart failure treatment.
Rehospitalization for heart failure until day 30 | 30 days
  Any visit to the hospital due to heart failure.
Death from all causes until day 30 | 30 days
Days alive out-of-intensive care unit until day 30 | 30 days
Renal replacement therapy until day 30 | 30 days
Quality of life at 30-day follow-up (5Q-DL) | 30 days
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Congestion assessed by Lung Ultrasound | 1 day
  Multiple b-lines in at least two windows (yes/no)
Time from inclusion to freedom from supplemental oxygen with a saturation >93% | Up to 30 days

OTHER OUTCOMES:
Pulmonary congestion on chest x-ray the next day | 1 day
Duration of index admission, including hospital-based rehabilitation | Up to 30 days
FiO2, Blood pressure, respiratory rate, heart rate after 1 hour | 1 hours
Echocardiographic parameters (LVEF, %) | After 24 hours after hospital-admission
NT-pro-BNP | After 24 hours after hospital-admission
  Measured and analysed at each site
Myocardial infarction within 48 hours | 2 days
  Assessed by the treating clinician
Change in bodyweight from baseline until 2 days (kg) | 2 days
  Measured at admission and after 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Grand, PhD, Principal Investigator — Hvidovre University Hospital
Locations (4):
- Denmark (4):
  - Bispebjerg Hospital, Copenhagen, Copenhagen
  - Hvidovre Hospital, Copenhagen, Copenhagen
  - Nordsjællands Hospital, Hillerød
  - Roskilde Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No